CLINICAL TRIAL: NCT04660253
Title: A Group Parenting Intervention for Depressed Fathers (LTP+ Dads): A Feasibility Study From Pakistan
Brief Title: Feasibility and Acceptability of Culturally Adapted Group Psychosocial Intervention for Depressed Fathers
Acronym: LTP-Dads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILL-Dads-001
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Long-Term Potentiation; amsonic acid

STUDY DESIGN:
Intervention Model Description: This integrated intervention is called LTP Plus Dads consisting of 10 group sessions delivered weekly by trained professionals who received weekly supervision by LTP Plus master trainers.
Masking Description: Researchers doing outcome assessments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LTP Plus Dads (Experimental): Participants in this group will receive 10 sessions of LTP plus dads
  Interventions: Behavioral: LTP Plus Dads

INTERVENTIONS:
Behavioral: LTP Plus Dads

SUMMARY:
The study is a feasibility trial with a pre and post-experiment design in Karachi, Pakistan's most populous city. The intervention comprises of twelve sessions of learning through play (LTP) plus during the three month period.

ELIGIBILITY:
Inclusion Criteria:

* Depressed fathers of children 0-30 months
* Given written informed consent

Exclusion Criteria:

* Not willing to participate
* Out of trial catchment area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Depressed Fathers of children 0-30 months
Enrollment: 18 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | Baseline to 3rd month
  Intervention feasibility tested by collating data on recruitment and retention rates. The success criterion of feasibility is to recruit > 50% of eligible fathers
Intervention acceptability | Baseline to 3rd month
  Intervention acceptability assessed using data on attendance. Criterion for acceptability is a mean attendance rate of >70% of at least 5 sessions.

SECONDARY OUTCOMES:
Change in severity of symptoms measured using Hamilton Depression Rating Scale (Hamilton, 1960) | Changes in severity of symptoms from baseline to 3rd month
  It is the most widely used clinician-administered depression assessment on a 3-point or 5-point Likert-type scale. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression; the maximum score being 52 on the 17-point scale
Changes in severity of symptoms measured using Edinburgh Postnatal Depression Scale (EPDS; Cox et al. 1987), | Changes in severity of symptoms from baseline to 3rd month
  A widely used 10-item measure of postnatal depression that has been used with fathers in the postnatal period. The higher score shows high severity of depression.

REFERENCES:
- [Derived] Husain MI, Chaudhry IB, Khoso AB, Wan MW, Kiran T, Shiri T, Chaudhry N, Mehmood N, Jafri SF, Naeem F, Husain N. A Group Parenting Intervention for Depressed Fathers (LTP + Dads): A Feasibility Study from Pakistan. Children (Basel). 2021 Jan 6;8(1):26. doi: 10.3390/children8010026. PMID 33419080